CLINICAL TRIAL: NCT01499277
Title: A Phase III, Multicentre, Randomised, Double-Blind Comparative Study to Evaluate the Efficacy and Safety of Ceftaroline Fosamil (600 mg Every 8 Hours) Versus Vancomycin Plus Aztreonam in the Treatment of Patients With Complicated Bacterial Skin and Soft Tissue Infections With Evidence of Systemic Inflammatory Response or Underlying Comorbidities
Brief Title: Evaluation of Ceftaroline Fosamil Versus Vancomycin Plus Aztreonam in the Treatment of Patients With Skin Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3720C00001; 2011-004013-16
Record Dates: First submitted 2011-12-16; First posted 2011-12-26 (Estimated); Results first posted 2015-11-09 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Complicated Skin and Soft Tissue Infection
Keywords: complicated skin and soft tissue infections (cSSTI); skin infection; ceftaroline; wound infection; cellulitis; burn infection; bacterial infection; vancomycin
MeSH Terms: conditions — Soft Tissue Infections; Cellulitis; Wound Infection; Bacterial Infections | interventions — Ceftaroline; Vancomycin; Aztreonam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Ceftaroline fosamil (Experimental): Patients will receive 600 mg of ceftaroline fosamil administered as a 120-minute intravenous infusion very 8 hours. Each dose will be infused in a volume of 250 mL over 120-minutes followed by aztreonam placebo in a volume of 100 mL infused over 30 minutes every 8 hours. In addition vancomycin placebo will be given in a volume of 250 mL infused over 120 minutes every 12 hours. Doses will be adjusted according to the patient's renal function.
  Interventions: Drug: Ceftaroline fosamil
- Vancomycin plus aztreonam (Active Comparator): Patients will receive combination of vancomycin plus aztreonam. Dose of vancomycin will be based on the patient's actual weight and will receive intravenous vancomycin every 12 hours with each dose infused over 120-minutes. Aztreonam dose will be 1 gram intravenously in a volume of 100 mL infused over 30 minutes every 8 hours. In addition, ceftaroline fosamil placebo will be given in a volume of 250 mL infused over 120 minutes every 8 hours. Doses adjusted according to patients renal function
  Interventions: Drug: Vancomycin; Drug: Aztreonam

INTERVENTIONS:
Drug: Ceftaroline fosamil — IV ceftaroline 600mg every 8 hours
  Arms: Ceftaroline fosamil
Drug: Vancomycin — IV vancomycin 15mg/kg every 12 hours
  Arms: Vancomycin plus aztreonam
Drug: Aztreonam — IV aztreonam 1 g every 8 hours
  Arms: Vancomycin plus aztreonam

SUMMARY:
The purpose of this study is to evaluate the effects of Ceftaroline Fosamil versus Vancomycin plus Aztreonam in treatment of patients with complicated bacterial skin and soft tissue infections.

DETAILED DESCRIPTION:
A Phase III, Multicentre, Randomised, Double-Blind Comparative Study to Evaluate the Efficacy and Safety of Ceftaroline Fosamil (600 mg every 8 hours) Versus Vancomycin Plus Aztreonam in the Treatment of Patients with Complicated Bacterial Skin and Soft Tissue Infections With Evidence of Systemic Inflammatory Response or Underlying Comorbidities

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years or older
* Complicated skin and skin structure infection (cSSTI)
* Infection of sufficient severity to warrant hospitalization
* Infection of sufficient severity such that it is expected to require at least 5 days of intravenous antibiotic therapy

Exclusion Criteria:

* Received systemic antibacterial drugs for greater than 24 hours within 96 hours prior to first dose of study drug
* Uncomplicated skin and skin structure infections, skin infections suspected to be caused by viral or fungal pathogens
* Diabetic foot infections, decubitus ulcers, ulcers due to peripheral vascular disease
* Infection caused by human or animal bites, sternal wound infections, bone infection or arthritis due to an infection, critical limb ischemia of the affected limb
* Chronic liver disease or severe impaired renal function, severe low white blood cell count, burns on greater than 15% of total body surface area, necrotizing skin infection, amputation required of primary site of infection, sustained shock

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 802 (Actual)
Dates: Start 2012-05; Primary Completion 2014-06 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Melnick, MSD, Study Director — AstraZeneca
Locations (91):
- United States (10):
  - Research Site, Chula Vista, California
  - Research Site, Orlando, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Carmel, Indiana
  - Research Site, Hazard, Kentucky
  - Research Site, Springfield, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Las Vegas, Nevada
  - Research Site, Garden City, New York
  - Research Site, Bellaire, Texas
- Argentina (2):
  - Research Site, Córdoba
  - Research Site, Santa Fe
- Research Site, Parkville, Australia
- Research Site, Brussels, Belgium
- Brazil (4):
  - Research Site, Belo Horizonte
  - Research Site, Passo Fundo
  - Research Site, Salvador
  - Research Site, São José do Rio Preto
- Bulgaria (3):
  - Research Site, Pleven
  - Research Site, Rousse
  - Research Site, Sofia
- Chile (2):
  - Research Site, Temuco
  - Research Site, Viña del Mar
- China (15):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Nanning
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shijiazhuang
  - Research Site, Wuhan
  - Research Site, Xi'an
- Croatia (2):
  - Research Site, Slavonski Brod
  - Research Site, Zagreb
- Czechia (2):
  - Research Site, Jihlava
  - Research Site, Pardubice
- Research Site, Orléans, France
- Germany (3):
  - Research Site, Dessau
  - Research Site, Hanau
  - Research Site, Heilbronn
- Research Site, Athens, Greece
- Hong Kong (2):
  - Research Site, Kowloon
  - Research Site, Pokfulam
- Israel (4):
  - Research Site, Haifa
  - Research Site, Ramat Gan
  - Research Site, Safed
  - Research Site, Tel Aviv
- Research Site, Milan, Italy
- Research Site, Guadalajara, Mexico
- Peru (2):
  - Research Site, Cusco
  - Research Site, Lima
- Philippines (2):
  - Research Site, Manila
  - Research Site, Quezon City
- Poland (2):
  - Research Site, Lodz
  - Research Site, Lublin
- Research Site, Bucharest, Romania
- Russia (6):
  - Research Site, Moscow
  - Research Site, Perm
  - Research Site, Saint Petersburg
  - Research Site, Smolensk
  - Research Site, Vsevolozhsk
  - Research Site, Yaroslavl
- South Africa (4):
  - Research Site, Benoni
  - Research Site, Cape Town
  - Research Site, Johannesburg
  - Research Site, Worcester
- South Korea (5):
  - Research Site, Ansan
  - Research Site, Deagu
  - Research Site, Incheon
  - Research Site, Seoul
  - Research Site, Wŏnju
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Granada
  - Research Site, Madrid
  - Research Site, Terrassa
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Taipei
  - Research Site, Yung Kang City
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Diyarbakır
  - Research Site, Izmir
- Ukraine (4):
  - Research Site, Cherkasy
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Odesa

REFERENCES:
- [Derived] Dryden M, Kantecki M, Yan JL, Stone GG, Leister-Tebbe H, Wilcox M. Treatment outcomes of secondary bacteraemia in patients treated with ceftaroline fosamil: pooled results from six phase III clinical trials. J Glob Antimicrob Resist. 2022 Mar;28:108-114. doi: 10.1016/j.jgar.2021.10.027. Epub 2021 Dec 16. PMID 34922058
- [Derived] Wilcox M, Yan JL, Gonzalez PL, Dryden M, Stone GG, Kantecki M. Impact of Underlying Comorbidities on Outcomes of Patients Treated with Ceftaroline Fosamil for Complicated Skin and Soft Tissue Infections: Pooled Results from Three Phase III Randomized Clinical Trials. Infect Dis Ther. 2022 Feb;11(1):217-230. doi: 10.1007/s40121-021-00557-w. Epub 2021 Nov 6. PMID 34741280
- [Derived] Sanchez-Garcia M, Hammond J, Yan JL, Kantecki M, Ansari W, Dryden M. Baseline Characteristics and Outcomes Among Patients with Complicated Skin and Soft Tissue Infections Admitted to the Intensive Care Unit: Analysis of the Phase 3 COVERS Randomized Trial of Ceftaroline Fosamil Versus Vancomycin Plus Aztreonam. Infect Dis Ther. 2020 Sep;9(3):609-623. doi: 10.1007/s40121-020-00297-3. Epub 2020 Jun 30. PMID 32607967
- [Derived] Corey GR, Wilcox MH, Gonzalez J, Jandourek A, Wilson DJ, Friedland HD, Das S, Iaconis J, Dryden M. Ceftaroline fosamil therapy in patients with acute bacterial skin and skin-structure infections with systemic inflammatory signs: A retrospective dose comparison across three pivotal trials. Int J Antimicrob Agents. 2019 Jun;53(6):830-837. doi: 10.1016/j.ijantimicag.2019.01.016. Epub 2019 Feb 1. PMID 30716446
- [Derived] Cheng K, Pypstra R, Yan JL, Hammond J. Summary of the safety and tolerability of two treatment regimens of ceftaroline fosamil: 600 mg every 8 h versus 600 mg every 12 h. J Antimicrob Chemother. 2019 Apr 1;74(4):1086-1091. doi: 10.1093/jac/dky519. PMID 30597021
- [Derived] Das S, Li J, Iaconis J, Zhou D, Stone GG, Yan JL, Melnick D. Ceftaroline fosamil doses and breakpoints for Staphylococcus aureus in complicated skin and soft tissue infections. J Antimicrob Chemother. 2019 Feb 1;74(2):425-431. doi: 10.1093/jac/dky439. PMID 30380060
- [Derived] Dryden M, Zhang Y, Wilson D, Iaconis JP, Gonzalez J. A Phase III, randomized, controlled, non-inferiority trial of ceftaroline fosamil 600 mg every 8 h versus vancomycin plus aztreonam in patients with complicated skin and soft tissue infection with systemic inflammatory response or underlying comorbidities. J Antimicrob Chemother. 2016 Dec;71(12):3575-3584. doi: 10.1093/jac/dkw333. Epub 2016 Sep 1. PMID 27585969

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 802 patients were enrolled from 111 centres in 6 regions in this study. The first patient was enrolled on 17 May 2012 and the last patient last visit was on 26 June 2014. Of 802 enrolled participants, 30 did not meet the eligibility criteria and 11 were randomized but not treated.
Groups:
- Ceftaroline: Ceftaroline fosamil at 600 mg every 8 hours (q8h)
- Vancomycin/Aztreonam: Vancomycin Plus Aztreonam
Period: Overall Study
Arm/Group | Ceftaroline | Vancomycin/Aztreonam
Started | 506 | 255
Completed | 459 | 223
Not Completed | 47 | 32
Not completed — Adverse Event | 3 | 6
Not completed — Death | 3 | 2
Not completed — Lost to Follow-up | 15 | 8
Not completed — Protocol Violation | 2 | 3
Not completed — Withdrawal by Subject | 16 | 6
Not completed — Lack of therapeutic response and other | 8 | 7

BASELINE CHARACTERISTICS:
Population: 761 randomized patients who received any amount of study therapy. there are 11 patients who are randomized , but didn't receive any study therapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceftaroline | Vancomycin/Aztreonam | Total
Number analyzed (Participants) | 506 | 255 | 761
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.6 (16.51) [18 to 91] | 53.6 (16.25) | 52.9 (16.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196 | 107 | 303
  Male | 310 | 148 | 458

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response at Test of Cure (TOC) in Modified Intent-to-treat (MITT) Analysis Set
Description: The observed difference in the clinical cure rates at TOC (ceftaroline group minus vancomycin plus aztreonam group) in MITT. Clinical cure rate is measured by comparing the participant's signs and symptoms at TOC visit to those recorded at study baseline.
Time Frame: 7 to 20 days after the last dose of study drug
Population: Modified intent-to-treat (MITT)
Measure: Number; unit: Participant
Arm/Group | Ceftaroline | Vancomycin/Aztreonam
Number analyzed (Participants) | 506 | 255
Participant
  Clinical cure | 396 [-6.9 to 5.41] | 202
  Clinical failure | 58 | 34
  indeterminate | 52 | 19
Statistical Analysis 1: Comparison: Ceftaroline vs Vancomycin/Aztreonam; The primary objective of this study was to determine the noninferiority in the clinical cure rate for ceftaroline compared vancomycin plus azreonam group at TOC in both MITT and CE populations; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI for the observed difference in the primary outcome measures (clinical cure rates) between ceftaroline group and vancomycin plus aztreonam group were calculated in both MITT and CE Populations at the TOC visit. Noninferiority was concluded if the lower limit of the 95% CI was higher than -10% in both MITT and CE Populations; RD is the difference in clinical cure rates (Ceftaroline minus Vancomycin/Aztreonam). CI was calculated by unstratified Miettinen and Nurminen CI; Risk Difference (RD) = -0.95, 95% CI 2-sided [-6.9 to 5.41] — CI for risk difference was estimated by 95% using unstratified Miettinen and Nurminen CI

2. Primary Outcome: Clinical Response at TOC in Clinically Evaluable (CE) Analysis Set
Description: The observed difference in the clinical cure rates at TOC (ceftaroline group minus vancomycin plus aztreonam group) in CE. Clinical cure rate is measured by comparing the participant's signs and symptoms at TOC visit to those recorded at study baseline.
Time Frame: 7 to 20 days after the last dose of study drug
Population: Clinical evaluable (CE)
Measure: Number; unit: Participant
Arm/Group | Ceftaroline | Vancomycin/Aztreonam
Number analyzed (Participants) | 395 | 211
Participant
  Clinical cure | 342 | 180
  Clinical failure | 53 | 31
Statistical Analysis 1: Comparison: Ceftaroline vs Vancomycin/Aztreonam; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI for the observed difference in the primary outcome measures (clinical cure rates) between ceftaroline group and vancomycin plus aztreonam group were calculated in both MITT and CE Populations at the TOC visit. Noninferiority was concluded if the lower limit of the 95% CI was higher than -10% in both MITT and CE Populations. If non-inferioirity was achieved then a test of superioirty was conducted if lower limit of 95% CI for the difference was >0%; RD is the difference in clinical cure rates (Ceftaroline minus Vancomycin/Aztreonam).CI was calculated by unstratified Miettinen and Nurminen CI; Risk Difference (RD) = 1.27, 95% CI 2-sided [-4.32 to 7.48] — CI for risk difference was estimated by 95% using unstratified Miettinen and Nurminen CI

3. Secondary Outcome: Per Patient Microbiological Response at TOC in Microbiologically Modified-intent-to-treat (mMITT) Analysis Set
Description: Difference in microbiological favorable response rate at TOC in mMITT analysis set. Favorable microbiological response rate is measured by comparing TOC microbiological data to baseline microbiological data. In the absence of TOC microbiological data it is presumed from the clinical response.
Time Frame: 7 to 20 days after the last dose of study drug
Population: Microbiologically modified-intent-to-treat (mMITT)
Measure: Number; unit: Participant
Arm/Group | Ceftaroline | Vancomycin/Aztreonam
Number analyzed (Participants) | 248 | 136
Participant
  Favorable | 203 | 109
  Unfavorable | 17 | 17
  Indeterminate | 28 | 10
Statistical Analysis 1: Comparison: Ceftaroline vs Vancomycin/Aztreonam; Test type: Superiority or Other; RD is the difference in favorable rates (Ceftaroline minus Vancomycin/Aztreonam).CI was calculated by unstratified Miettinen and Nurminen CI; Risk Difference (RD) = 1.71, 95% CI 2-sided [-6.21 to 10.39] — CI for risk difference was estimated by 95% using unstratified Miettinen and Nurminen CI

4. Secondary Outcome: Per-patient Micro Response at TOC in Microbiologically Evaluable (ME) Analysis Set
Description: Difference in microbiological favorable response rate at TOC in ME. Favourable microbiological response rate is measured by comparing TOC microbiological data to baseline microbiological data. In the absence of TOC microbiological data it is presumed from the clinical response.
Time Frame: 7 to 20 days after the last dose of study drug
Population: Microbiologically evaluable (ME)
Measure: Number; unit: Participant
Arm/Group | Ceftaroline | Vancomycin/Aztreonam
Number analyzed (Participants) | 181 | 112
Participant
  Favourable | 167 | 98
  Unfavorable | 14 | 14
Statistical Analysis 1: Comparison: Ceftaroline vs Vancomycin/Aztreonam; Test type: Superiority or Other; [statistical method as in outcome 3, analysis 1]; Risk Difference (RD) = 4.77, 95% CI 2-sided [-2.11 to 12.86] — CI for risk difference was estimated by 95% using unstratified Miettinen and Nurminen CI

5. Secondary Outcome: Clinical Response at End of Treatment (EOT) in MITT Analysis Set
Description: The observed difference in the clinical cure rates at EOT (ceftaroline group minus vancomycin plus aztreonam group) in MITT. Clinical cure rate is measured by comparing the participant's signs and symptoms at EOT visit to those recorded at study baseline.
Time Frame: On day of last dose of study drug (or + 1 day)
Measure: Number; unit: Participants
Arm/Group | Ceftaroline | Vancomycin/Aztreonam
Number analyzed (Participants) | 506 | 255
Participants
  Clinical cure | 429 | 213
  Clinical failure | 44 | 29
  Indeterminate | 31 | 11
  Missing | 2 | 2
Statistical Analysis 1: Comparison: Ceftaroline vs Vancomycin/Aztreonam; Test type: Superiority or Other; RD is the difference in cure rates (Ceftaroline minus Vancomycin/Aztreonam).CI was calculated by unstratified Miettinen and Nurminen CI; Risk Difference (RD) = 1.25, 95% CI 2-sided [-4.05 to 7.06] — CI for risk difference was estimated by 95% using unstratified Miettinen and Nurminen CI

6. Secondary Outcome: Clinical Response at EOT in CE Analysis Set
Description: The observed difference in the clinical cure rates at EOT (ceftaroline group minus vancomycin plus aztreonam group) in CE. Clinical cure rate is measured by comparing the participant's signs and symptoms at EOT visit to those recorded at study baseline.
Time Frame: On day of last dose of study drug (or +1 day)
Measure: Number; unit: Participants
Arm/Group | Ceftaroline | Vancomycin/Aztreonam
Number analyzed (Participants) | 395 | 211
Participants
  Clinical cure | 356 | 184
  Clinical failure | 39 | 27
Statistical Analysis 1: Comparison: Ceftaroline vs Vancomycin/Aztreonam; Test type: Superiority or Other; [statistical method as in outcome 5, analysis 1]; Risk Difference (RD) = 2.92, 95% CI 2-sided [-2.19 to 8.73] — CI for risk difference was estimated by 95% using unstratified Miettinen and Nurminen CI

7. Secondary Outcome: Clinical Relapse at Late Follow-up (LFU) in CE Patients Who Were Cured at TOC
Description: The observed difference in the clinical relapse rates at LFU (ceftaroline group minus vancomycin plus aztreonam group) in CE. Clinical relapse rate at LFU is measured by comparing a patient's signs and symptoms at late follow-up to those when they were cured at TOC.
Time Frame: 21 to 42 days after the last dose of study drug
Measure: Number; unit: Participants
Arm/Group | Ceftaroline | Vancomycin/Aztreonam
Number analyzed (Participants) | 342 | 180
Participants
  Relapse | 3 | 3
  No relapse | 335 | 174
  Indeterminate | 3 | 3
  Missing | 1 | 0
Statistical Analysis 1: Comparison: Ceftaroline vs Vancomycin/Aztreonam; Test type: Superiority or Other; RD is the difference in relapse rates (Ceftaroline minus Vancomycin/Aztreonam).CI was calculated by unstratified Miettinen and Nurminen CI; Risk Difference (RD) = -0.79, 95% CI 2-sided [-3.98 to 1.18] — CI for risk difference was estimated by 95% using unstratified Miettinen and Nurminen CI

8. Secondary Outcome: Early Response at 48 to 72 Hours of Treatment in MITT Analysis Set
Description: The observed difference in the early success rates at 48 to 72 hours of treatment (ceftaroline group minus vancomycin plus aztreonam group) in MITT. Early response rate as measured by comparing the participant's signs and symptoms at the 48-72 hour visit to those recorded at study baseline.
Time Frame: 48 to 72 hours after first dose of study drug
Measure: Number; unit: Participants
Arm/Group | Ceftaroline | Vancomycin/Aztreonam
Number analyzed (Participants) | 506 | 255
Participants
  success | 445 | 229
  failure | 28 | 11
  Indeterminate | 33 | 15
Statistical Analysis 1: Comparison: Ceftaroline vs Vancomycin/Aztreonam; Test type: Superiority or Other; RD is the difference in success rates (Ceftaroline minus Vancomycin/Aztreonam).CI was calculated by unstratified Miettinen and Nurminen CI; Risk Difference (RD) = -1.86, 95% CI 2-sided [-6.34 to 3.15] — CI for risk difference was estimated by 95% using unstratified Miettinen and Nurminen CI

9. Secondary Outcome: Per-pathogen Microbiological Response at TOC by Baseline Pathogen From Site of Skin Infection in ME
Description: Per-pathogen microbiological response at TOC by baseline pathogen from site of skin infection in ME analysis set
Time Frame: 7 to 20 days after the last dose of study drug
Measure: Number; unit: Participants
Arm/Group | Ceftaroline | Vancomycin/Aztreonam
Number analyzed (Participants) | 181 | 112
Participants
  MSSA - Favorable; (n=94, 57) | 91 | 49
  MSSA - Unfavorable; (n=94, 57) | 3 | 8
  MRSA - Favorable; (n=25, 15) | 22 | 12
  MRSA - Unfavorable; (n=25, 15) | 3 | 3
  Streptococcus pyogenes - Favorable; (n=15, 7) | 14 | 7
  Streptococcus pyogenes - Unfavorable; (n=15, 7) | 1 | 0
  Streptococcus agalactiae - Favorable; (n=6, 9) | 6 | 9
  Streptococcus agalactiae - Unfavorable; (n=6, 9) | 0 | 0
  Streptococcus dysgalactiae - Favorable; (n=9, 0) | 9 | 0
  Streptococcus dysgalactiae - Unfavorable; (n=9, 0) | 0 | 0
  Enterococcus faecalis - Favorable; (n=6, 5) | 5 | 4
  Enterococcus faecalis - Unfavorable; (n=6, 5) | 1 | 1
  Escherichia coli - Favorable; (n=12, 10) | 12 | 9
  Escherichia coli - Unfavorable; (n=12, 10) | 0 | 1
  Klebsiella pneumoniae - Favorable; (n=7, 4) | 6 | 3
  Klebsiella pneumoniae - Unfavorable; (n=7, 4) | 1 | 1
  Klebsiella oxytoca - Favorable; (n=4, 1) | 4 | 1
  Klebsiella oxytoca - Unfavorable; (n=4, 1) | 0 | 0
  Proteus mirabilis - Favorable; (n=7, 2) | 6 | 2
  Proteus mirabilis - Unfavorable; (n=7, 2) | 1 | 0
  Morganella morganii - Favorable; (n=4, 2) | 4 | 2
  Morganella morganii - Unfavorable; (n=4, 2) | 0 | 0
  Enterobacter cloacae - Favorable; (n=4, 5) | 4 | 5
  Enterobacter cloacae - Unfavorable; (n=4, 5) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of the first dose of study drug up to TOC visit (8 to 15 days after the last dose). Serious AEs were collected from time of signature of informed consent up to the LFU visit (21 to 35 days after the last dose).
Arm/Group | Ceftaroline | Vancomycin/Aztreonam
Serious Adverse Events (participants affected / at risk) | 31/506 | 15/255
Other Adverse Events (participants affected / at risk) | 82/506 | 46/255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ceftaroline (N=506) | Vancomycin/Aztreonam (N=255)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Diabetic gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Metal poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0/0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1/1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary haemosiderosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftaroline (N=506) | Vancomycin/Aztreonam (N=255)
Anaemia (Blood and lymphatic system disorders) | 10 (10) | 9 (9)
Constipation (Gastrointestinal disorders) | 9 (9) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 12 (12) | 5 (5)
Nausea (Gastrointestinal disorders) | 20 (20) | 11 (11)
Vomiting (Gastrointestinal disorders) | 13 (15) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 14 (14) | 8 (9)
Headache (Nervous system disorders) | 17 (17) | 12 (13)
Rash (Skin and subcutaneous tissue disorders) | 10 (11) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to use such Confidential study information and not to disclose them to any other third parties, except that the undersigned shall not be prevented from using or disclosing information: (a) which by written records was previously known; (b) which is now public knowledge, (c) which is lawfully obtained by the undersigned from sources who have a lawful right to disclose such information.